CLINICAL TRIAL: NCT02069795
Title: Utilization of Speech Analysis as a Diagnostic Tool to Objectively Evaluate Early Signs of Mild Traumatic Brain Injury: A Pilot Study
Brief Title: Speech Analysis as a Diagnostic Tool for Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forte Sports Medicine and Orthopedics (Other)
Collaborators: Waveform Communications LLC (Unknown)
Responsible Party: Principal Investigator, Terry G Horner, Physician, Forte Sports Medicine and Orthopedics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB # 1312958125
Record Dates: First submitted 2014-02-17; First posted 2014-02-24 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Concussion
Keywords: concussion, athlete, speech analysis
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Voice recording (Experimental): Subjects voices were recorded as they spoke specific words
  Interventions: Other: Voice recording

INTERVENTIONS:
Other: Voice recording

SUMMARY:
The waveform assessment of an athlete's speech production has a high probability of showing abnormalities after brain injury (concussions) which could be used not only for diagnosis of the concussion, but for recovery of the brain. The aim of this study is to investigate this possibility using the Cobweb automated application system for acoustic processing.

DETAILED DESCRIPTION:
Concussions affect cognitive and fine muscle motor control, and these changes will be reflected in the acoustic characteristics of the vowels being produced. The methods to identify and analyze the acoustics of vowels will greatly extend the detailed understanding of vowels produced after a concussion. The identification of the changes in formant frequencies, pitch, and duration will provide the means to use these parameters as an automated diagnostic tool. The waveform assessment of the athlete's speech production has a high probability of showing brain abnormalities immediately after a suspected or diagnosed concussion at the venue of the athletic sport. The aim of this study assessment is to investigate this possibility using the Cobweb system and greatly enhance the ability to diagnose a concussion in a timely manner to remove the athlete from practice or play.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed or suspected of having a sports concussion seen in a clinical setting
* Ages 6 -21

Exclusion Criteria:

* Patients who have physical injuries to their lips, tongue or oral cavity will be excluded until they have healed.
* Patients with hearing or speech abnormalities who cannot consistently produce the stimulus materials.
* Non-native speakers who cannot read the materials or produce the stimuli consistently.
* Patients who cannot read the materials or produce the stimuli consistently due to their age.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in formant frequencies | 2 months
  1. Changes in formant frequencies F0,F1,F2,F3 in patients following concussion to recovery time.

SECONDARY OUTCOMES:
Changes in duration of speech production | 2 months
  Changes in duration of speech production in patients following concussion to recovery time .

CONTACTS AND LOCATIONS:
Overall Officials: Terry G Horner, MD, Principal Investigator — Forte Sports Medicine and Orthopedics